CLINICAL TRIAL: NCT02376907
Title: Multinational Study on Endoscopic Management of Distal Malignant Biliary Obstruction Combined With Gastric Outlet Obstruction
Brief Title: Biliary Drainage in Patients With Duodenal Metal Stent
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Hiroyuki Isayama, MD, PhD, Associate Professor, Tokyo University
Other Study IDs: 10639
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Jaundice
Keywords: distal malignant biliary obstruction; endoscopic retrograde cholangiopancreatography; endoscopic ultrasound; gastric outlet obstruction; stent
MeSH Terms: conditions — Jaundice; Gastric Outlet Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EUS-BD or ERCP with duodenal SEMS: Patients who underwent endoscopic placement of a duodenal self-expandable metal stent (SEMS) for nonresectable malignant GOO and endoscopic biliary drainage for nonresectable distal MBO.
  Interventions: Procedure: Biliary drainage

INTERVENTIONS:
Procedure: Biliary drainage — EUS-BD or ERCP

SUMMARY:
This is a retrospective study to evaluate the outcomes of endoscopic biliary drainage according to the timing of distal malignant biliary obstruction (MBO) in relation to gastric outlet obstruction (GOO) and the location of GOO.

DETAILED DESCRIPTION:
This is a multinational multicenter retrospective cohort study to evaluate the outcomes of endoscopic biliary drainage in patients with a duodenal SEMS. Endoscopic ultrasound-guided biliary drainage (EUS-BD), including choledochoduodenostomy, hepaticogastrostomy, antegrade biliary stenting or a combination, and endoscopic retrograde cholangiopancreatography (ERCP) with stenting are to be compared. Specifically, the outcomes are to be evaluated according to the timing of distal MBO in relation to GOO and the location of GOO.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic placement of a duodenal SEMS for nonresectable malignant GOO.
* Patients who underwent endoscopic biliary drainage for nonresectable MBO.
* MBO was located ≥ 2 cm from the bifurcation.
* Patients who could be followed up more than three months after completion of both biliary drainage and duodenal SEMS placement.
* Age ≥20 years.
* Irrespective of sex and a primary disease.

Exclusion Criteria:

* Patients who underwent surgical bypass for GOO.
* Patients who underwent percutaneous and surgical biliary drainage prior to the placement of duodenal SEMS.
* Patients with altered gastrointestinal anatomy (Billroth-II reconstruction, Roux-en-Y reconstruction, etc.).
* Patients who would not give a consent to the report of their own data.
* Patients considered ineligible for inclusion in the study by an investigator for other reasons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent the initial duodenal SEMS between Jan/1/2010 and Jun/30/2014 are included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time to recurrent biliary obstruction | Up to 1 year
  Recurrent biliary obstruction is defined as a composite endpoint of either occlusion or migration of biliary stent, and time to recurrent biliary obstruction is time from biliary drainage to recurrence of biliary obstruction.

SECONDARY OUTCOMES:
Causes of recurrent biliary obstruction | Up to 1 year
  Causes of recurrent biliary obstruction include sludge, food impaction, ingrowth, tumor overgrowth, hemobilia and others.
Functional success rate of biliary drainage | 2 weeks
  Functional success is defined when bilirubin decreases < 50% or is normalized within 2 weeks.
Procedure-related complication of biliary drainage and duodenal meta stent placement (type and severity) | 30 days
  Complications and their severity are determined using the American Society of Gastrointestinal Endoscopy guidelines.
Survival time | Up to 2 year
  Survival time is defined as the period between biliary stent placement and death.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Isayama, MD, PhD, Principal Investigator — Graduate School of Medicine, The University of Tokyo
Locations (25):
- Eastern Hepatobiliary Hospital, Second Military Medical University, Shanghai, China
- The Prince of Wales Hospital, Shatin, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, India
- Japan (14):
  - Fukushima Medical University, Fukushima
  - Gifu University, Gifu
  - Onomichi General Hospital, Hiroshima
  - Teine-Keijinkai Hospital, Hokkaido
  - Sapporo Medical University, Hokkaido
  - Hokkaido University School of Medicine, Hokkaido
  - Kinki University, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Graduate School of Medicine, The University of Tokyo, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
  - Kanto Central Hospital, Tokyo
  - Tokyo Medical University, Tokyo
  - Tokyo Metropolitan Police Hospital, Tokyo
- Prince Court Medical Center, Kuala Lumpur, Malaysia
- Singapore (2):
  - Singapore General Hospital, Outram Road
  - Changi General Hospital, Simei New Town
- South Korea (2):
  - Asan Medical Center, Seoul
  - Soon Chun Hyang University School of Medicine, Seoul
- National Taiwan University Hospital, Taipei, Taiwan
- Thailand (2):
  - Chulalongkorn University, Bangkok
  - Rajavithi Hospital, Bangkok

REFERENCES:
- [Background] Maire F, Hammel P, Ponsot P, Aubert A, O'Toole D, Hentic O, Levy P, Ruszniewski P. Long-term outcome of biliary and duodenal stents in palliative treatment of patients with unresectable adenocarcinoma of the head of pancreas. Am J Gastroenterol. 2006 Apr;101(4):735-42. doi: 10.1111/j.1572-0241.2006.00559.x. PMID 16635221
- [Background] Kaw M, Singh S, Gagneja H. Clinical outcome of simultaneous self-expandable metal stents for palliation of malignant biliary and duodenal obstruction. Surg Endosc. 2003 Mar;17(3):457-61. doi: 10.1007/s00464-002-8541-3. Epub 2002 Oct 31. PMID 12404053
- [Background] Mutignani M, Tringali A, Shah SG, Perri V, Familiari P, Iacopini F, Spada C, Costamagna G. Combined endoscopic stent insertion in malignant biliary and duodenal obstruction. Endoscopy. 2007 May;39(5):440-7. doi: 10.1055/s-2007-966327. PMID 17516351
- [Background] Moon JH, Choi HJ. Endoscopic double-metallic stenting for malignant biliary and duodenal obstructions. J Hepatobiliary Pancreat Sci. 2011 Sep;18(5):658-63. doi: 10.1007/s00534-011-0409-2. PMID 21655973
- [Background] Hamada T, Nakai Y, Isayama H, Sasaki T, Kogure H, Kawakubo K, Sasahira N, Yamamoto N, Togawa O, Mizuno S, Ito Y, Hirano K, Toda N, Tada M, Koike K. Duodenal metal stent placement is a risk factor for biliary metal stent dysfunction: an analysis using a time-dependent covariate. Surg Endosc. 2013 Apr;27(4):1243-8. doi: 10.1007/s00464-012-2585-9. Epub 2012 Oct 17. PMID 23073685
- [Background] Kahaleh M, Hernandez AJ, Tokar J, Adams RB, Shami VM, Yeaton P. Interventional EUS-guided cholangiography: evaluation of a technique in evolution. Gastrointest Endosc. 2006 Jul;64(1):52-9. doi: 10.1016/j.gie.2006.01.063. PMID 16813803
- [Background] Horaguchi J, Fujita N, Noda Y, Kobayashi G, Ito K, Obana T, Takasawa O, Koshita S, Kanno Y. Endosonography-guided biliary drainage in cases with difficult transpapillary endoscopic biliary drainage. Dig Endosc. 2009 Oct;21(4):239-44. doi: 10.1111/j.1443-1661.2009.00899.x. PMID 19961522
- [Background] Itoi T, Isayama H, Sofuni A, Itokawa F, Kurihara T, Tsuchiya T, Tsuji S, Ishii K, Ikeuchi N, Tanaka R, Umeda J, Moriyasu F, Kawakami H. Stent selection and tips on placement technique of EUS-guided biliary drainage: transduodenal and transgastric stenting. J Hepatobiliary Pancreat Sci. 2011 Sep;18(5):664-72. doi: 10.1007/s00534-011-0410-9. PMID 21688214
- [Background] Kawakubo K, Isayama H, Nakai Y, Sasahira N, Kogure H, Sasaki T, Hirano K, Tada M, Koike K. Simultaneous Duodenal Metal Stent Placement and EUS-Guided Choledochoduodenostomy for Unresectable Pancreatic Cancer. Gut Liver. 2012 Jul;6(3):399-402. doi: 10.5009/gnl.2012.6.3.399. Epub 2012 Jul 12. PMID 22844572
- [Derived] Hamada T, Nakai Y, Lau JY, Moon JH, Hayashi T, Yasuda I, Hu B, Seo DW, Kawakami H, Kuwatani M, Katanuma A, Kitano M, Ryozawa S, Hanada K, Iwashita T, Ito Y, Yagioka H, Togawa O, Maetani I, Isayama H. International study of endoscopic management of distal malignant biliary obstruction combined with duodenal obstruction. Scand J Gastroenterol. 2018 Jan;53(1):46-55. doi: 10.1080/00365521.2017.1382567. Epub 2017 Oct 6. PMID 28982258
- See also: Tokyo Conference of Asian Pancreato-biliary Interventional Endoscopist — http://www.t-cap.jp/